CLINICAL TRIAL: NCT03718390
Title: A Multicentre, Randomised, Controlled, Observer-Blind Study to Evaluate Safety and Gastric Retention Properties of Modified Release Prototype Capsules (LYN-PLT) in Healthy Adults
Brief Title: Study to Evaluate Safety/Duration in Stomach of Extended Release Capsules in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lyndra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LYN-PLT-C-001; ACTRN12618000991213 (Registry Identifier: ANZCTR); CM8818 (Other: CMAX)
Record Dates: First submitted 2018-10-14; First posted 2018-10-24 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Gastric Retention; Healthy
MeSH Terms: interventions — D-Worm; Granuflex E; Endoscopy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: A total of 40 eligible subjects participate in the Dosing and Observation period. The enrollment occurs in five Dosing Groups. Within each Dosing Group, subjects are randomized to receive either one of four LYN-PLT extended release capsules or a placebo capsule (8 per formulation).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing simple randomization via computerized sequence generation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sentinel Group 1 LYN-PLT (Experimental): Sentinel dosing in endoscopy center of one of each formulation (A, B, C, D, E) in a 1:1:1:1:1 ratio (centralized randomized, observer blind) and evaluation of gastric retention by MRI
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Procedure: Endoscopy; Procedure: Magnetic Resonance Imaging
- Sentinel Group 2 LYN-PLT (Experimental): Sentinel dosing (second) in endoscopy center of one of each formulation (A, B, C, D, E) in a 1:1:1:1:1 ratio (centralized randomized, observer blind) and evaluation of gastric retention by MRI
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Procedure: Endoscopy; Procedure: Magnetic Resonance Imaging
- Group 3 LYN-PLT (Experimental): Dosing in clinic of two of each formulation (A, B, C, D, E) in a 1:1:1:1:1 ratio (centralized, randomized, observer blind). and evaluation of gastric retention by MRI
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Procedure: Magnetic Resonance Imaging
- Group 4 LYN-PLT (Experimental): Dosing in clinic of two of each formulation (A, B, C, D, E) in a 1:1:1:1:1 ratio (centralized, randomized, observer blind) and evaluation of gastric retention by MRI
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Procedure: Magnetic Resonance Imaging
- Group 5 LYN-PLT (Experimental): Dosing in clinic of two of each formulation (A, B, C, D, E) in a 1:1:1:1:1 ratio (centralized, randomized, observer blind) and evaluation of gastric retention by MRI.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Formulation A — Formulation A (37/40A) of LYN-PLT containing less than 300 mg sucrose within the extended release formulation
  Other Names: LYN-PLT Formulation A
Drug: Formulation B — Formulation B (46/40A) of LYN-PLT containing less than 300 mg sucrose within the extended release formulation
  Other Names: LYN-PLT Formulation B
Drug: Formulation C — Formulation C (37/50A) of LYN-PLT containing less than 300 mg sucrose within the extended release formulation
  Other Names: LYN-PLT Formulation C
Drug: Formulation D — Formulation D (46/50A) of LYN-PLT containing less than 300 mg sucrose within the extended release formulation
  Other Names: LYN-PLT Formulation D
Drug: Formulation E — Placebo Capsule containing microcrystalline cellulose
  Other Names: Placebo capsule
Procedure: Endoscopy — Endoscopy at 2 hours post dosing
  Arms: Sentinel Group 1 LYN-PLT; Sentinel Group 2 LYN-PLT
Procedure: Magnetic Resonance Imaging — MRI will be performed on specified days according to protocol
  Other Names: MRI

SUMMARY:
To assess how long extended release prototype capsule formulations stay in the stomach as determined by magnetic resonance imaging (MRI).

To evaluate the safety of several extended release capsule formulations (LYN-PLT) and a placebo capsule.

DETAILED DESCRIPTION:
This is a multicentre, observer blind, randomised, single dose study in healthy adult subjects.

The first 5 subjects enrolled into the study will be regarded as Dosing Group 1 (sentinel group) and assigned to each of the five available study formulations. Dosing of subjects in Dosing Groups 1 and 2 will be performed at the endoscopy centre. Dosing of subjects in Dosing Groups 3 through 5 will be performed at the clinical site.

Subjects remain in the inpatient unit for 7 days after dosing. During this time, subjects undergo intermittent imaging assessments for gastric retention (MRI and abdominal U/S), safety assessments and faecal collections for assessments of retrieved components and bowel movement characteristics.

Subjects return to the clinic on Days 10, 15, 22 and 29 (End of Study visit). Safety assessments will be performed at all visits. MRI, abdominal U/S and outpatient faecal collections may continue based on the clinical findings from subjects dosed with modified release capsule formulations. On Day 29, the subjects will undergo final safety assessments at the clinic and thereafter, will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects
2. Body mass index of 18.0 to 30.0 kg/meters-squared
3. Suitable scores for two swallowing questionnaires
4. Demonstrate normal swallowing and gastrointestinal passage for capsule, as assessed while undergoing imaging studies
5. Must provide written informed consent

Exclusion Criteria:

1. Participants who have previously been enrolled in this study
2. History of any drug or alcohol abuse in the past 2 years
3. Current smokers and those who have smoked within the past 12 months
4. Individuals with clinically significant medical history relating to the gastrointestinal tract and potential complications, thereof
5. Individuals with a positive test for HIV, hepatitis B or hepatitis C
6. Serious adverse reaction or serious hypersensitivity to components of the study formulations or patency capsule
7. Individuals who have received any experimental agent within 30 days (or 5 half-lives), whichever is longer, prior to the date of dosing
8. Individuals with contraindication to MRI imaging
9. Individuals with functional constipation, irritable bowel, or functional diarrhea, as evaluated by standardized questionnaire
10. Individuals with contraindications to elective X-ray based on known or expected radiation exposure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Gastric retention assessed by Magnetic Resonance Imaging (MRI) | Up to 9 Days post-dosing
  Visualization of formulation/formulation components in the stomach by MRI
Safety and tolerability of four LYN-PLT modified release capsules and a placebo capsule collected from Adverse Event (AE) reporting based on spontaneous reports | Through study completion, up to 6 months
  The number of confirmed gastrointestinal adverse events will be reported based on spontaneous adverse event reporting
Safety and tolerability of four LYN-PLT modified release capsules and a placebo capsule collected from Adverse Event (AE) reporting based on changes in examinations pre (Day 1) and post dosing (Days 4 and 7) | Through study completion, up to 6 months
  Clinically significant aggregate changes in vital signs, physical examinations and safety laboratory assessments (haematology, liver function tests, clinical chemistry panel) between pre-dose (Day 1) and post-dosing (Day 4 and 7) will be reported as AE's
Safety and tolerability of four LYN-PLT modified release capsules and a placebo capsule collected from Adverse Event (AE) reporting based on post dosing evaluation of bowel movements for blood | Through study completion, up to 6 months
  Examination and reporting of post-dosing bowel movements for blood; clinically significant abnormal findings will be reported as AE's.
Safety and tolerability of four LYN-PLT modified release capsules and a placebo capsule collected from Adverse Event (AE) reporting | Through study completion, up to 6 months
  If abdominal pain occurs, a systematic algorithm to evaluate abdominal pain [modified Structured Assessment of GastroIntestinal Symptoms (SAGIS)] will be used. Clinically significantly abnormal findings will be reported as adverse events

SECONDARY OUTCOMES:
Gastric retention assessed by abdominal ultrasound (U/S) | Up to 9 Days post-dosing
  Visualization of formulation/formulation components in the stomach by U/S
Confirm esophageal clearance of several MR capsules and a placebo capsule | 2 hours post dosing
  For Group 1 and Group 2 via endoscopy
Physical Feature of Recovered Formulation Components | Through study completion up to Day 29
  Record the physical features, e.g. number of polymeric arms (if separate) or if attached to the core, of formulation components recovered from collected fecal specimens

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No